CLINICAL TRIAL: NCT02675452
Title: A Phase 1 First in Human Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 176 in Subjects With Relapsed or Refractory Multiple Myeloma and Subjects With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: AMG 176 First in Human Trial in Participants With Relapsed or Refractory Multiple Myeloma and Participants With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: sponsor decision, unrelated to safety
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150161; 2015-004777-32 (EudraCT Number)
Record Dates: First submitted 2015-12-22; First posted 2016-02-05 (Estimated); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Relapsed or Refractory Multiple Myeloma; Relapsed or Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Recurrence; Multiple Myeloma; Leukemia, Myeloid, Acute | interventions — tapotoclax; Azacitidine; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- AMG 176 - Part 1a (Experimental): Part 1a - Participants with muliple myeloma (MM) administered AMG 176 as an intravenous (IV) infusion for two-consecutive days (QD2) followed by a 5 days break.
  Interventions: Drug: AMG 176
- AMG 176 - Part 1b (Experimental): Part 1b - Participants with multiple myeloma (MM) administered AMG 176 as an intravenous (IV) infusion, once a week (QW) followed by 6 days break.
  Interventions: Drug: AMG 176
- AMG 176 - Part 3a (Experimental): Part 3a - Participants with acute myeloid leukemia (AML) administered AMG 176 as an intravenous (IV) infusion once a day, for two-consecutive days (QD2) followed by a 5 day break.
  Interventions: Drug: AMG 176
- AMG 176 - Part 3b (Experimental): Part 3b - Participants with acute myeloid leukemia (AML) administered AMG 176 as an intravenous (IV) infusion, once a week (QW) followed by 6 days break.
  Interventions: Drug: AMG 176
- AMG 176 - Part 3c (Experimental): Part 3c - Participants in Japan only with acute myeloid leukemia (AML) administered AMG 176 as an intravenous (IV) infusion, once a week (QW) followed by 6 days break.
  Interventions: Drug: AMG 176
- AMG 176 - Part 3d (Experimental): Part 3d - Participants in the United States with acute myeloid leukemia (AML) administered AMG 176 as an intravenous (IV) infusion, once a week (QW), for 3 weeks, in combination with itraconazole.
  Interventions: Drug: AMG 176; Drug: Itraconazole
- AMG 176 - Part 4 (Experimental): Part 4 - Participants with acute myeloid leukemia (AML) administered AMG 176 as an intravenous (IV) infusion, either once a week (QW) followed by 6 days break, or once a day, for two-consecutive days (QD2), in combination with azacitidine.
  Interventions: Drug: AMG 176; Drug: Azacitidine
- AMG 176 - Part 5 (Experimental): Part 5 - Participants with acute myeloid leukemia (AML) administered AMG 176 as an intravenous (IV) infusion at the maximum tolerated combination dose from Part 4, either once a week (QW) followed by 6 days break, or once a day, for two-consecutive days (QD2), in combination with azacitidine.
  Interventions: Drug: AMG 176; Drug: Azacitidine

INTERVENTIONS:
Drug: AMG 176 — Study Drug
  Other Names: Study Investigational Product (IP)
Drug: Azacitidine — Non-investigational product
  Arms: AMG 176 - Part 4; AMG 176 - Part 5
Drug: Itraconazole — Non-investigational product
  Arms: AMG 176 - Part 3d

SUMMARY:
The main objectives are to evaluate the safety and tolerability of AMG 176 monotherapy in participants with relapsed or refractory multiple myeloma and participants with relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
This is a Phase 1, first-in-human, multicenter; non-randomized, open-label and dose-exploration study of AMG 176 administered IV in participants with relapsed or refractory multiple myeloma and participants with relapsed or refractory acute myeloid leukemia The study will be conducted in five parts.

ELIGIBILITY:
INCLUSION CRITERIA:

* For participants in Japan only: if a participant is younger than 20 years at the time of signing the informed consent form, informed consent must be obtained from both the participant and his/her legal representative
* (Multiple myeloma [MM] participants) Pathologically documented, multiple myeloma relapsed or refractory disease after at least 2 lines of therapy
* (MM participants only) Measurable disease per the International Myeloma Working Group response criteria
* (Acute myeloid leukemia [AML] participants) AML as defined by the World Health Organization Classification persisting or recurring following one or more treatment courses, and for participants in Japan, determined by the investigator to be not eligible for approved anticancer drug therapy in Japan; EXCEPT acute promyelocytic leukemia.
* (AML participants only) More than 5% blasts in bone marrow and Circulating white blood cells < 25,000/ul.
* Must be willing and able to undergo a core bone marrow biopsy (MM participants only) and bone marrow aspirate (MM and AML participants) at screening.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2,
* (MM partiicpants only) Satisfactory hematological function without transfusion or growth factor support
* Life expectancy of > 3 months, in the opinion of the investigator
* Adequate hepatic function
* Adequate cardiac function
* Adequate renal function
* Female participants of childbearing potential must have a negative serum or urine pregnancy test
* Other inclusion criteria may apply

EXCLUSION CRITERIA:

* Previously received an allogeneic stem cell transplant within 6 months OR having received immunosuppressive therapy within the last three months OR having signs or symptoms of acute or chronic graft-versus-host disease
* Autologous stem cell transplant less than 90 days prior to study day 1
* (MM participants only) MM with Immunoglobulin M subtype
* (MM participants only) Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal protein, Skin changes syndrome
* (MM participants only) Existing plasma cell leukemia
* (MM participants only) Waldenstrom's macroglobulinemia
* (MM participants only) Amyloidosis
* Infection requiring intravenous anti-infective treatments within 1 week of study enrollment (day 1)
* Myocardial infarction within 6 months of enrollment, symptomatic congestive heart failure (New York Heart Association > class II)
* History of arterial thrombosis (eg, stroke or transient ischemic attack) in the past 6 months prior to enrollment
* Currently receiving treatment in another investigational device or drug study. Other investigational procedures while participating in this study will be allowed if approved by Amgen medical monitor
* Participants with elevated cardiac troponin above the manufacturer's 99th percentile upper reference limit for ADVIA Centaur XP assay at screening performed by the central laboratory
* Participants with evidence of recent cardiac injury at screening based on creatine kinase-muscle/brain, N-terminal prohormone of brain natriuretic peptide, and electrocardiogram
* Other exclusion criteria may apply
* (AML Part 3d only) History of QT prolongation, torsades de pointes, ventricular tachycardia and cardiac arrest
* History or evidence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection unless agreed upon with medical monitor.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (24):
- United States (10):
  - City of Hope National Medical Center, Duarte, California
  - University of California Davis Medical Center, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - Northside Hospital, Atlanta, Georgia
  - University of Chicago Hospital, Chicago, Illinois
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (3):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Canada (2):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - University Health Network-Princess Margaret Cancer Centre, Toronto, Ontario
- Germany (4):
  - Universitaetsklinikum der Rheinisch-Westfaelischen Technischen Hochschule Aachen, Aachen
  - Universitaetsklinikum Bonn, Bonn
  - Universitaetsklinikum Ulm, Ulm
  - Universitaetsklinikum Wuerzburg, Würzburg
- Japan (5):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - National Hospital Organization Okayama Medical Center, Okayama, Okayama-ken
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 21 study centers in the United States, Canada, Australia, Germany, and Japan, and participated from June 2016 to May 2024. The study was conducted in multiple parts and Part 5 did not enroll any participants due to early termination of the study. Part 2 was removed during a protocol amendment.
Pre-assignment Details: Participants with multiple myeloma (MM) or with acute myeloid leukemia (AML) were enrolled into 29 cohorts. Dosing of AMG 176 was from Dose A (lowest) to Dose I (highest).
Groups:
- Part 1A Cohort 1 (MM): AMG 176 Dose A Twice Weekly (BIW): Participants with MM received AMG 176 Dose A BIW. AMG 176 was administered as an intravenous (IV) infusion in a 4-week cycle.
- Part 1A Cohort 2 (MM): AMG 176 Dose B BIW: Participants with MM received AMG 176 Dose B IV BIW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 1A Cohort 3 (MM): AMG 176 Dose C BIW: Participants with MM received AMG 176 Dose C BIW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 1A Cohort 4 (MM): AMG 176 Dose D BIW: Participants with MM received AMG 176 Dose D BIW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 1A Cohort 5 (MM): AMG 176 Dose E BIW: Participants with MM received AMG 176 Dose E BIW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 1A Cohort 6 (MM): AMG 176 Dose G BIW: Participants with MM received AMG 176 Dose G BIW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 1A Cohort 7 (MM): AMG 176 Dose E Then Dose F BIW: Participants with MM received AMG 176 Dose E in cycle 1 week 1, then received Dose F BIW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 1A Cohort 8 (MM): AMG 176 Dose E Then Dose G BIW: Participants with MM received AMG 176 Dose E in cycle 1 week 1, then received Dose G BIW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 1A Cohort 9 (MM): AMG 176 Dose E Then Dose H BIW: Participants with MM received AMG 176 Dose E in cycle 1 week 1, then received Dose H BIW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 1A Cohort 10 (MM): AMG 176 Dose E Then Dose I BIW: Participants with MM received AMG 176 Dose E in cycle 1 week 1, then received Dose I BIW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 1B Cohort 1 (MM): AMG 176 Dose E Then Dose F Once Weekly (QW): Participants with MM received AMG 176 Dose E in cycle 1 week 1, then received Dose F QW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 1B Cohort 2 (MM): AMG 176 Dose E Then Dose G QW: Participants with MM received AMG 176 Dose E in cycle 1 week 1, then received Dose G QW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 1B Cohort 3 (MM): AMG 176 Dose E Then Dose H QW: Participants with MM received AMG 176 Dose E in cycle 1 week 1, then received Dose H QW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 1B Cohort 4 (MM): AMG 176 Dose E Then Dose I QW: Participants with MM received AMG 176 Dose E in cycle 1 week 1, then received Dose I QW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 3A Cohort 1 (AML): AMG 176 Dose D BIW: Participants with AML received AMG 176 Dose D BIW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 3A Cohort 2 (AML): AMG 176 Dose E BIW: Participants with AML received AMG 176 Dose E BIW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 3A Cohort 3 (AML): AMG 176 Dose E Then Dose F BIW: Participants with AML received AMG 176 Dose E in cycle 1 week 1, then received Dose F BIW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 3A Cohort 4 (Japanese Participants With AML): AMG 176 Dose E Then Dose F QW: Japanese participants with AML received AMG 176 Dose E in cycle 1 week 1, then received Dose F QW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 3B Cohort 1 (AML): AMG 176 Dose E QW: Participants with AML received AMG 176 Dose E QW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 3B Cohort 2 (AML): AMG 176 Dose E Then Dose F QW: Participants with AML received AMG 176 Dose E in cycle 1 week 1, then received Dose F QW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 3B Cohort 3 (AML): AMG 176 Dose E Then Dose G QW: Participants with AML received AMG 176 Dose E in cycle 1 week 1, then received Dose G QW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 3C Cohort 1 (Japanese Participants With AML): AMG 176 Dose E QW: Japanese participants with AML received AMG 176 Dose E QW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 3D Cohort 1 (AML): AMG 176 Dose D QW + Itraconazole: Participants with AML received AMG 176 Dose D QW. AMG 176 was administered as an IV infusion in a 4-week cycle. They also received 200 mg itraconazole once daily (QD) for 7 days in week 1.
- Part 4 Cohort 1 (AML): AMG 176 Dose D QW + Azacitidine: Participants with AML received AMG 176 Dose D QW. AMG 176 was administered as an IV infusion in a 4-week cycle. They also received 75 mg/m^2 azacitidine subcutaneously (SC) or IV QD for 7 days in week 1.
- Part 4 Cohort 2 (AML): AMG 176 Dose E QW + Azacitidine: Participants with AML received AMG 176 Dose E QW. AMG 176 was administered as an IV infusion in a 4-week cycle. They also received 75 mg/m^2 azacitidine SC or IV QD for 7 days in week 1.
- Part 4 Cohort 3 (AML): AMG 176 Dose E Then Dose F QW + Azacitidine: Participants with AML received AMG 176 Dose E in cycle 1 week 1, then received Dose F QW. AMG 176 was administered as an IV infusion in a 4-week cycle. They also received 75 mg/m^2 azacitidine SC or IV QD for 7 days in week 1.
- Part 4 Cohort 4 (AML): AMG 176 Dose E Then Dose G QW + Azacitidine: Participants with AML received AMG 176 Dose E in cycle 1 week 1, then received Dose G QW. AMG 176 was administered as an IV infusion in a 4-week cycle. They also received 75 mg/m^2 azacitidine SC or IV QD for the first 7 days of the 4-week cycle.
- Part 4 Cohort 5A (AML): AMG 176 Dose E BIW + Azacitidine: Participants with AML received AMG 176 Dose E BIW. AMG 176 was administered as an IV infusion in a 4-week cycle. They also received 75 mg/m^2 azacitidine SC or IV QD for the first 7 days of the 4-week cycle.
- Part 4 Cohort 5B (AML): AMG 176 Dose E the Dose G BIW + Azacitidine: Participants with AML received AMG 176 Dose E in cycle 1 week 1, then received Dose G BIW. AMG 176 was administered as an IV infusion in a 4-week cycle. They also received 75 mg/m^2 azacitidine SC or IV QD for the first 7 days of the 4-week cycle.
Period: Overall Study
Arm/Group | Part 1A Cohort 1 (MM): AMG 176 Dose A Twice Weekly (BIW) | Part 1A Cohort 2 (MM): AMG 176 Dose B BIW | Part 1A Cohort 3 (MM): AMG 176 Dose C BIW | Part 1A Cohort 4 (MM): AMG 176 Dose D BIW | Part 1A Cohort 5 (MM): AMG 176 Dose E BIW | Part 1A Cohort 6 (MM): AMG 176 Dose G BIW | Part 1A Cohort 7 (MM): AMG 176 Dose E Then Dose F BIW | Part 1A Cohort 8 (MM): AMG 176 Dose E Then Dose G BIW | Part 1A Cohort 9 (MM): AMG 176 Dose E Then Dose H BIW | Part 1A Cohort 10 (MM): AMG 176 Dose E Then Dose I BIW | Part 1B Cohort 1 (MM): AMG 176 Dose E Then Dose F Once Weekly (QW) | Part 1B Cohort 2 (MM): AMG 176 Dose E Then Dose G QW | Part 1B Cohort 3 (MM): AMG 176 Dose E Then Dose H QW | Part 1B Cohort 4 (MM): AMG 176 Dose E Then Dose I QW | Part 3A Cohort 1 (AML): AMG 176 Dose D BIW | Part 3A Cohort 2 (AML): AMG 176 Dose E BIW | Part 3A Cohort 3 (AML): AMG 176 Dose E Then Dose F BIW | Part 3A Cohort 4 (Japanese Participants With AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 1 (AML): AMG 176 Dose E QW | Part 3B Cohort 2 (AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 3 (AML): AMG 176 Dose E Then Dose G QW | Part 3C Cohort 1 (Japanese Participants With AML): AMG 176 Dose E QW | Part 3D Cohort 1 (AML): AMG 176 Dose D QW + Itraconazole | Part 4 Cohort 1 (AML): AMG 176 Dose D QW + Azacitidine | Part 4 Cohort 2 (AML): AMG 176 Dose E QW + Azacitidine | Part 4 Cohort 3 (AML): AMG 176 Dose E Then Dose F QW + Azacitidine | Part 4 Cohort 4 (AML): AMG 176 Dose E Then Dose G QW + Azacitidine | Part 4 Cohort 5A (AML): AMG 176 Dose E BIW + Azacitidine | Part 4 Cohort 5B (AML): AMG 176 Dose E the Dose G BIW + Azacitidine
Started | 3 | 3 | 4 | 3 | 3 | 2 | 4 | 4 | 5 | 5 | 3 | 3 | 3 | 3 | 6 | 5 | 5 | 2 | 4 | 3 | 4 | 4 | 10 | 5 | 5 | 4 | 13 | 10 | 13
Received AMG 176 | 3 | 3 | 4 | 3 | 3 | 2 | 4 | 4 | 5 | 5 | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 2 | 4 | 3 | 4 | 4 | 10 | 5 | 4 | 4 | 13 | 10 | 13
Completed | 3 | 2 | 3 | 3 | 3 | 1 | 4 | 4 | 4 | 3 | 3 | 2 | 1 | 0 | 4 | 3 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not Completed | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 3 | 2 | 2 | 3 | 0 | 4 | 3 | 3 | 3 | 10 | 5 | 4 | 4 | 12 | 9 | 13
Not completed — Sponsor decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 3 | 4
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 4 | 3 | 3 | 3 | 7 | 5 | 3 | 4 | 7 | 6 | 9
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who received at least 1 dose of AMG 176.
Groups:
- Part 1A Cohort 1 (MM): AMG 176 Dose A BIW: Participants with MM received AMG 176 Dose A BIW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 1B Cohort 1 (MM): AMG 176 Dose E Then Dose F QW: Participants with MM received AMG 176 Dose E in cycle 1 week 1, then received Dose F QW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 3D Cohort 1 (AML): AMG 176 Dose D QW + Itraconazole: Participants with AML received AMG 176 Dose D QW. AMG 176 was administered as an IV infusion in a 4-week cycle. They also received 200 mg itraconazole QD for 7 days in week 1.
- Part 4 Cohort 1 (AML): AMG 176 Dose D QW + Azacitidine: Participants with AML received AMG 176 Dose D QW. AMG 176 was administered as an IV infusion in a 4-week cycle. They also received 75 mg/m^2 azacitidine SC or IV QD for 7 days in week 1.
- Part 4 Cohort 4 (AML): AMG 176 Dose E Then Dose G QW + Azacitidine: Participants with AML received AMG 176 Dose E in cycle 1 week 1, then received Dose G QW. AMG 176 was administered as an IV infusion in a 4-week cycle. They also received 75 mg/m^2 azacitidine SC or IV QD for 7 days in week 1.
- Part 4 Cohort 5A (AML): AMG 176 Dose E BIW + Azacitidine: Participants with AML received AMG 176 Dose E BIW. AMG 176 was administered as an IV infusion in a 4-week cycle. They also received 75 mg/m^2 azacitidine SC or IV QD for 7 days in week 1.
- Part 4 Cohort 5B (AML): AMG 176 Dose E the Dose G BIW + Azacitidine: Participants with AML received AMG 176 Dose E in cycle 1 week 1, then received Dose G BIW. AMG 176 was administered as an IV infusion in a 4-week cycle. They also received 75 mg/m^2 azacitidine SC or IV QD for 7 days in week 1.
- Total: Total of all reporting groups
Arm/Group | Part 1A Cohort 1 (MM): AMG 176 Dose A BIW | Part 1A Cohort 2 (MM): AMG 176 Dose B BIW | Part 1A Cohort 3 (MM): AMG 176 Dose C BIW | Part 1A Cohort 4 (MM): AMG 176 Dose D BIW | Part 1A Cohort 5 (MM): AMG 176 Dose E BIW | Part 1A Cohort 6 (MM): AMG 176 Dose G BIW | Part 1A Cohort 7 (MM): AMG 176 Dose E Then Dose F BIW | Part 1A Cohort 8 (MM): AMG 176 Dose E Then Dose G BIW | Part 1A Cohort 9 (MM): AMG 176 Dose E Then Dose H BIW | Part 1A Cohort 10 (MM): AMG 176 Dose E Then Dose I BIW | Part 1B Cohort 1 (MM): AMG 176 Dose E Then Dose F QW | Part 1B Cohort 2 (MM): AMG 176 Dose E Then Dose G QW | Part 1B Cohort 3 (MM): AMG 176 Dose E Then Dose H QW | Part 1B Cohort 4 (MM): AMG 176 Dose E Then Dose I QW | Part 3A Cohort 1 (AML): AMG 176 Dose D BIW | Part 3A Cohort 2 (AML): AMG 176 Dose E BIW | Part 3A Cohort 3 (AML): AMG 176 Dose E Then Dose F BIW | Part 3A Cohort 4 (Japanese Participants With AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 1 (AML): AMG 176 Dose E QW | Part 3B Cohort 2 (AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 3 (AML): AMG 176 Dose E Then Dose G QW | Part 3C Cohort 1 (Japanese Participants With AML): AMG 176 Dose E QW | Part 3D Cohort 1 (AML): AMG 176 Dose D QW + Itraconazole | Part 4 Cohort 1 (AML): AMG 176 Dose D QW + Azacitidine | Part 4 Cohort 2 (AML): AMG 176 Dose E QW + Azacitidine | Part 4 Cohort 3 (AML): AMG 176 Dose E Then Dose F QW + Azacitidine | Part 4 Cohort 4 (AML): AMG 176 Dose E Then Dose G QW + Azacitidine | Part 4 Cohort 5A (AML): AMG 176 Dose E BIW + Azacitidine | Part 4 Cohort 5B (AML): AMG 176 Dose E the Dose G BIW + Azacitidine | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 2 | 4 | 4 | 5 | 5 | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 2 | 4 | 3 | 4 | 4 | 10 | 5 | 4 | 4 | 13 | 10 | 13 | 139
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 2 | 2 | 3 | 1 | 1 | 1 | 2 | 2 | 1 | 2 | 1 | 1 | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 3 | 4 | 2 | 4 | 2 | 0 | 4 | 3 | 4 | 51
  65 - 74 years | 1 | 1 | 0 | 1 | 2 | 0 | 2 | 1 | 4 | 3 | 2 | 2 | 1 | 2 | 1 | 3 | 2 | 1 | 2 | 1 | 0 | 0 | 5 | 0 | 1 | 1 | 6 | 5 | 3 | 53
  75 - 84 years | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 3 | 1 | 1 | 3 | 3 | 2 | 5 | 33
  >=85 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2 | 0 | 0 | 3 | 1 | 2 | 1 | 2 | 2 | 2 | 0 | 4 | 0 | 4 | 2 | 0 | 2 | 1 | 2 | 3 | 0 | 1 | 1 | 3 | 4 | 6 | 50
  Male | 2 | 3 | 3 | 1 | 3 | 2 | 1 | 3 | 3 | 4 | 1 | 1 | 1 | 3 | 1 | 5 | 1 | 0 | 4 | 1 | 3 | 2 | 7 | 5 | 3 | 3 | 10 | 6 | 7 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 10
  Not Hispanic or Latino | 3 | 3 | 4 | 3 | 3 | 2 | 3 | 4 | 4 | 5 | 3 | 3 | 3 | 3 | 4 | 5 | 5 | 2 | 4 | 3 | 2 | 4 | 7 | 3 | 4 | 4 | 12 | 10 | 13 | 128
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 1 | 6 | 4 | 19
  Black or African American | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 3 | 3 | 3 | 2 | 3 | 2 | 4 | 4 | 4 | 4 | 2 | 2 | 3 | 2 | 4 | 4 | 5 | 0 | 3 | 2 | 3 | 0 | 8 | 5 | 4 | 4 | 11 | 4 | 9 | 107
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5

OUTCOME MEASURES:

1. Secondary Outcome: Best Overall Response According to Revised International Working Group Uniform Response Criteria (IMWG-URC) for MM Participants (Parts 1A and 1B)
Description: A response consisted of any of the following, assessed according to the IMWG-URC: stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), minor response (MR), stable disease (SD), or progressive disease (PD) per IMWG-URC. CR: negative immunofixation on serum and urine, soft tissue plasmacytomas disappearance, < 5% plasma cells in bone marrow (BM). sCR: CR and normal serum free light chain ratio and no clonal cells in BM by immunohistochemistry. VGPR: Serum and urine M-protein detectable by immunofixation or ≥ 90% reduction in serum M-protein (urine M-protein level < 100 mg/24-hrs). PR: ≥ 50% reduction of serum M-protein and reduction in 24-hrs urinary M-protein by ≥ 90% or to < 200 mg/24-hours; MR: 25-49% reduction in serum M-protein and 50-89% reduction in 24-hr urinary M-protein (>200 mg/24-hrs); SD: not meeting criteria for CR, VGPR, PR, or PD; PD: ≥ 25% increase in serum or urine M-component, BM plasma cell percentages.
Time Frame: Day 1 cycle 1 to end of study; median duration from start of study treatment to end of study for all participants was 2.2 months
Population: The FAS included all participants who received at least 1 dose of AMG 176.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Cohort 1 (MM): AMG 176 Dose A BIW | Part 1A Cohort 2 (MM): AMG 176 Dose B BIW | Part 1A Cohort 3 (MM): AMG 176 Dose C BIW | Part 1A Cohort 4 (MM): AMG 176 Dose D BIW | Part 1A Cohort 5 (MM): AMG 176 Dose E BIW | Part 1A Cohort 6 (MM): AMG 176 Dose G BIW | Part 1A Cohort 7 (MM): AMG 176 Dose E Then Dose F BIW | Part 1A Cohort 8 (MM): AMG 176 Dose E Then Dose G BIW | Part 1A Cohort 9 (MM): AMG 176 Dose E Then Dose H BIW | Part 1A Cohort 10 (MM): AMG 176 Dose E Then Dose I BIW | Part 1B Cohort 1 (MM): AMG 176 Dose E Then Dose F QW | Part 1B Cohort 2 (MM): AMG 176 Dose E Then Dose G QW | Part 1B Cohort 3 (MM): AMG 176 Dose E Then Dose H QW | Part 1B Cohort 4 (MM): AMG 176 Dose E Then Dose I QW
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 2 | 4 | 4 | 5 | 5 | 3 | 3 | 3 | 3
Participants
  sCR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VGPR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  MR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SD | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
  PD | 3 | 3 | 4 | 2 | 3 | 1 | 4 | 3 | 2 | 5 | 3 | 1 | 1 | 3
  No post-baseline response evaluation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0

2. Secondary Outcome: Best Overall Response According to the 2017 European LeukemiaNet (ELN) Criteria in AML Participants (Parts 3A, 3B, 3C, 3D, and 4)
Description: A response was of any of the following, per the ELN criteria: Complete remission (CR) without minimal residual disease (CRMRD-), CR, CR with incomplete hematology recovery (CRi), morphologic leukemia-free state (MLFS), partial remission (PR), SD, PD. CRMRD-: CR with negativity for genetic marker by quantitative reverse transcription (RT-qPCR) or multicolor flow cytometry (MFC); CR: BM blasts <5% bone marrow, no circulating blasts/ extramedullary disease, ANC > 1.0 x 10^9/L, platelets ≥ 100 x 10^9/L; CRi: CR except for neutropenia (< 1.0 x 10^9/L) or thrombocytopenia (< 100 x 10^9/L); MLFS: BM blasts < 5% no blasts with auer rods/extramedullary disease, no hematologic recovery; PR: hematological criteria of CR; decrease BM blast to 5-25%; decrease of BM blast percentage by ≤ 50%; SD: absence of CRMRD-, CR, CRi, PR, MLFS and criteria for PD not met; PD: evidence of increase in BM blast percentage and/or increase of absolute blast count.
Time Frame: as for outcome 1
Population: The FAS included all participants who received at least 1 dose of AMG 176.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3A Cohort 1 (AML): AMG 176 Dose D BIW | Part 3A Cohort 2 (AML): AMG 176 Dose E BIW | Part 3A Cohort 3 (AML): AMG 176 Dose E Then Dose F BIW | Part 3A Cohort 4 (Japanese Participants With AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 1 (AML): AMG 176 Dose E QW | Part 3B Cohort 2 (AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 3 (AML): AMG 176 Dose E Then Dose G QW | Part 3C Cohort 1 (Japanese Participants With AML): AMG 176 Dose E QW | Part 3D Cohort 1 (AML): AMG 176 Dose D QW + Itraconazole | Part 4 Cohort 1 (AML): AMG 176 Dose D QW + Azacitidine | Part 4 Cohort 2 (AML): AMG 176 Dose E QW + Azacitidine | Part 4 Cohort 3 (AML): AMG 176 Dose E Then Dose F QW + Azacitidine | Part 4 Cohort 4 (AML): AMG 176 Dose E Then Dose G QW + Azacitidine | Part 4 Cohort 5A (AML): AMG 176 Dose E BIW + Azacitidine | Part 4 Cohort 5B (AML): AMG 176 Dose E the Dose G BIW + Azacitidine
Number analyzed (Participants) | 5 | 5 | 5 | 2 | 4 | 3 | 4 | 4 | 10 | 5 | 4 | 4 | 13 | 10 | 13
Participants
  CRMRD- | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
  CRi | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  MLFS | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
  PR | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SD | 1 | 0 | 0 | 1 | 3 | 2 | 1 | 1 | 3 | 2 | 3 | 3 | 5 | 5 | 7
  PD | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  No post-baseline response evaluation | 2 | 4 | 3 | 1 | 0 | 0 | 2 | 2 | 7 | 3 | 0 | 0 | 3 | 3 | 5

3. Primary Outcome: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT)
Description: A DLT was assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v 4.0, and considered by the investigators to be related to AMG 176. A DLT was defined as a grade 3 or higher non-hematological or a grade 4 hematologic adverse event (AE) that occurred during the DLT observation period.
  CTCAE is graded from grade 1 to 5, with higher grades indicating a worse outcome, and included; grade 1 = mild, grade 2= moderate, grade 3 = severe, grade 4 = life-threatening, and grade 5 = death.
Time Frame: Days 1 to 28 of cycle 1 (4 weeks)
Population: DLT-evaluable analysis set included participants if they experienced a DLT during the DLT evaluation period or if they received at least 75% of the planned doses of AMG 176 (and 100% of the planned doses of azacitidine in Part 4) and completed the DLT evaluation period.
Measure: Count of Participants; unit: Participants
Groups:
- Part 4 Cohort 5B (AML): AMG 176 Dose E the Dose G BIW + Azacitidine: Participants with AML received AMG 176 Dose E in cycle 1 week 1, then received Dose G BIW. AMG 176 was administered as an IV infusion in a 4-week cycle. They also received 75 mg/m^2 azacitidine SC or IV QD for for 7 days in week 1.
Arm/Group | Part 1A Cohort 1 (MM): AMG 176 Dose A BIW | Part 1A Cohort 2 (MM): AMG 176 Dose B BIW | Part 1A Cohort 3 (MM): AMG 176 Dose C BIW | Part 1A Cohort 4 (MM): AMG 176 Dose D BIW | Part 1A Cohort 5 (MM): AMG 176 Dose E BIW | Part 1A Cohort 6 (MM): AMG 176 Dose G BIW | Part 1A Cohort 7 (MM): AMG 176 Dose E Then Dose F BIW | Part 1A Cohort 8 (MM): AMG 176 Dose E Then Dose G BIW | Part 1A Cohort 9 (MM): AMG 176 Dose E Then Dose H BIW | Part 1A Cohort 10 (MM): AMG 176 Dose E Then Dose I BIW | Part 1B Cohort 1 (MM): AMG 176 Dose E Then Dose F QW | Part 1B Cohort 2 (MM): AMG 176 Dose E Then Dose G QW | Part 1B Cohort 3 (MM): AMG 176 Dose E Then Dose H QW | Part 1B Cohort 4 (MM): AMG 176 Dose E Then Dose I QW | Part 3A Cohort 1 (AML): AMG 176 Dose D BIW | Part 3A Cohort 2 (AML): AMG 176 Dose E BIW | Part 3A Cohort 3 (AML): AMG 176 Dose E Then Dose F BIW | Part 3A Cohort 4 (Japanese Participants With AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 1 (AML): AMG 176 Dose E QW | Part 3B Cohort 2 (AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 3 (AML): AMG 176 Dose E Then Dose G QW | Part 3C Cohort 1 (Japanese Participants With AML): AMG 176 Dose E QW | Part 3D Cohort 1 (AML): AMG 176 Dose D QW + Itraconazole | Part 4 Cohort 1 (AML): AMG 176 Dose D QW + Azacitidine | Part 4 Cohort 2 (AML): AMG 176 Dose E QW + Azacitidine | Part 4 Cohort 3 (AML): AMG 176 Dose E Then Dose F QW + Azacitidine | Part 4 Cohort 4 (AML): AMG 176 Dose E Then Dose G QW + Azacitidine | Part 4 Cohort 5A (AML): AMG 176 Dose E BIW + Azacitidine | Part 4 Cohort 5B (AML): AMG 176 Dose E the Dose G BIW + Azacitidine
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 2 | 4 | 4 | 5 | 5 | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 2 | 4 | 3 | 4 | 4 | 10 | 5 | 4 | 4 | 13 | 10 | 13
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

4. Primary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a clinical trial participant.
  A TEAE was an AE that started on or after the first dose of investigational product (AMG 176) up to 30 days after the end of investigational product. Any clinically significant changes in vital signs, electrocardiograms, and clinical laboratory tests were reported as TEAEs.
  A treatment-related AE was any TEAE that per investigator review had a reasonable possibility of being caused by the investigational product (AMG 176).
Time Frame: Day 1 cycle 1 to 30 days after the last dose of AMG 176; median treatment duration was 1.2 months
Population: The FAS included all participants that received at least 1 dose of AMG 176.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Cohort 1 (MM): AMG 176 Dose A BIW | Part 1A Cohort 2 (MM): AMG 176 Dose B BIW | Part 1A Cohort 3 (MM): AMG 176 Dose C BIW | Part 1A Cohort 4 (MM): AMG 176 Dose D BIW | Part 1A Cohort 5 (MM): AMG 176 Dose E BIW | Part 1A Cohort 6 (MM): AMG 176 Dose G BIW | Part 1A Cohort 7 (MM): AMG 176 Dose E Then Dose F BIW | Part 1A Cohort 8 (MM): AMG 176 Dose E Then Dose G BIW | Part 1A Cohort 9 (MM): AMG 176 Dose E Then Dose H BIW | Part 1A Cohort 10 (MM): AMG 176 Dose E Then Dose I BIW | Part 1B Cohort 1 (MM): AMG 176 Dose E Then Dose F QW | Part 1B Cohort 2 (MM): AMG 176 Dose E Then Dose G QW | Part 1B Cohort 3 (MM): AMG 176 Dose E Then Dose H QW | Part 1B Cohort 4 (MM): AMG 176 Dose E Then Dose I QW | Part 3A Cohort 1 (AML): AMG 176 Dose D BIW | Part 3A Cohort 2 (AML): AMG 176 Dose E BIW | Part 3A Cohort 3 (AML): AMG 176 Dose E Then Dose F BIW | Part 3A Cohort 4 (Japanese Participants With AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 1 (AML): AMG 176 Dose E QW | Part 3B Cohort 2 (AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 3 (AML): AMG 176 Dose E Then Dose G QW | Part 3C Cohort 1 (Japanese Participants With AML): AMG 176 Dose E QW | Part 3D Cohort 1 (AML): AMG 176 Dose D QW + Itraconazole | Part 4 Cohort 1 (AML): AMG 176 Dose D QW + Azacitidine | Part 4 Cohort 2 (AML): AMG 176 Dose E QW + Azacitidine | Part 4 Cohort 3 (AML): AMG 176 Dose E Then Dose F QW + Azacitidine | Part 4 Cohort 4 (AML): AMG 176 Dose E Then Dose G QW + Azacitidine | Part 4 Cohort 5A (AML): AMG 176 Dose E BIW + Azacitidine | Part 4 Cohort 5B (AML): AMG 176 Dose E the Dose G BIW + Azacitidine
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 2 | 4 | 4 | 5 | 5 | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 2 | 4 | 3 | 4 | 4 | 10 | 5 | 4 | 4 | 13 | 10 | 13
Participants
  TEAEs | 3 | 2 | 4 | 3 | 3 | 2 | 4 | 4 | 5 | 5 | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 2 | 4 | 3 | 4 | 4 | 10 | 5 | 4 | 4 | 13 | 10 | 13
  Treatment-related TEAEs | 2 | 1 | 3 | 3 | 3 | 2 | 3 | 2 | 5 | 5 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 2 | 2 | 3 | 2 | 3 | 5 | 5 | 4 | 4 | 11 | 8 | 8

5. Primary Outcome: Maximum Observed Concentration (Cmax) of AMG 176
Description: Plasma concentrations of AMG 176 were determined using a validated assay. Noncompartmental analysis was performed for estimation of pharmacokinetic (PK) parameters. Concentrations below the lower limit of quantification (LLOQ) of 5.00 ng/mL were set to zero before data analysis.
Time Frame: Parts 1B, 3B, 3C, 3A (cohort 4) Cycle 1: day 1 pre, end of infusion (EOI), 1, 2, 3, 5, 7 hrs EOI, day 8 pre, EOI; Part 3D also days 9, 15 pre and EOI; Parts 1A, 3 (except cohort 4), 4: also day 2 pre, EOI, 1, 2, 3, 5, 7 hrs EOI, day 9 pre and EOI
Population: The PK analysis set included all participants who had received at least 1 dose of AMG 176 and had at least 1 PK sample collected. Participants with data available at each time point are presented.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Part 1A Cohort 1 (MM): AMG 176 Dose A BIW | Part 1A Cohort 2 (MM): AMG 176 Dose B BIW | Part 1A Cohort 3 (MM): AMG 176 Dose C BIW | Part 1A Cohort 4 (MM): AMG 176 Dose D BIW | Part 1A Cohort 5 (MM): AMG 176 Dose E BIW | Part 1A Cohort 6 (MM): AMG 176 Dose G BIW | Part 1A Cohort 7 (MM): AMG 176 Dose E Then Dose F BIW | Part 1A Cohort 8 (MM): AMG 176 Dose E Then Dose G BIW | Part 1A Cohort 9 (MM): AMG 176 Dose E Then Dose H BIW | Part 1A Cohort 10 (MM): AMG 176 Dose E Then Dose I BIW | Part 1B Cohort 1 (MM): AMG 176 Dose E Then Dose F QW | Part 1B Cohort 2 (MM): AMG 176 Dose E Then Dose G QW | Part 1B Cohort 3 (MM): AMG 176 Dose E Then Dose H QW | Part 1B Cohort 4 (MM): AMG 176 Dose E Then Dose I QW | Part 3A Cohort 1 (AML): AMG 176 Dose D BIW | Part 3A Cohort 2 (AML): AMG 176 Dose E BIW | Part 3A Cohort 3 (AML): AMG 176 Dose E Then Dose F BIW | Part 3A Cohort 4 (Japanese Participants With AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 1 (AML): AMG 176 Dose E QW | Part 3B Cohort 2 (AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 3 (AML): AMG 176 Dose E Then Dose G QW | Part 3C Cohort 1 (Japanese Participants With AML): AMG 176 Dose E QW | Part 3D Cohort 1 (AML): AMG 176 Dose D QW + Itraconazole | Part 4 Cohort 1 (AML): AMG 176 Dose D QW + Azacitidine | Part 4 Cohort 2 (AML): AMG 176 Dose E QW + Azacitidine | Part 4 Cohort 3 (AML): AMG 176 Dose E Then Dose F QW + Azacitidine | Part 4 Cohort 4 (AML): AMG 176 Dose E Then Dose G QW + Azacitidine | Part 4 Cohort 5A (AML): AMG 176 Dose E BIW + Azacitidine | Part 4 Cohort 5B (AML): AMG 176 Dose E the Dose G BIW + Azacitidine
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 2 | 3 | 4 | 5 | 5 | 3 | 3 | 2 | 3 | 5 | 5 | 5 | 2 | 4 | 3 | 4 | 4 | 9 | 0 | 0 | 0 | 0 | 10 | 13
ng/mL
  Cycle 1 day 1: number analyzed (Participants) | 3 | 3 | 4 | 2 | 3 | 2 | 3 | 2 | 4 | 3 | 3 | 3 | 2 | 2 | 5 | 5 | 5 | 2 | 4 | 3 | 4 | 4 | 9 | 0 | 0 | 0 | 0 | 10 | 13
  Cycle 1 day 1 | 2270 [1980 to 3690] | 2900 [1730 to 4340] | 3590 [1490 to 4310] | 5790 [4420 to 7160] | 10100 [9640 to 19000] | 26100 [25500 to 26700] | 10100 [7490 to 14200] | 24700 [3180 to 46200] | 4880 [3580 to 5920] | 5440 [3950 to 8590] | 7940 [7010 to 9760] | 6450 [6390 to 7460] | 12100 [3080 to 21100] | 4590 [4130 to 5050] | 5140 [3000 to 11900] | 5570 [3260 to 13800] | 6250 [4010 to 30800] | 7790 [7400 to 8180] | 3600 [2850 to 5880] | 5230 [3070 to 5360] | 3270 [0.00 to 5510] | 6290 [5900 to 7210] | 1670 [0.00 to 2400] |  |  |  |  | 5500 [0.00 to 21900] | 5380 [0.00 to 10700]
  Cycle 1 day 2: number analyzed (Participants) | 3 | 3 | 4 | 2 | 3 | 1 | 3 | 4 | 5 | 5 | 0 | 0 | 0 | 0 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 11
  Cycle 1 day 2 | 1780 [1490 to 4080] | 3800 [2340 to 5420] | 3570 [1290 to 4910] | 8270 [7020 to 9520] | 11800 [11200 to 12900] | 27300 [27300 to 27300] | 6500 [2890 to 8400] | 7980 [6770 to 42600] | 5230 [0.00 to 16600] | 7670 [4590 to 32000] |  |  |  |  | 6280 [2760 to 16100] | 7250 [4620 to 21600] | 6910 [4340 to 128000] |  |  |  |  |  |  |  |  |  |  | 4200 [0.00 to 23500] | 7050 [3440 to 143000]
  Cycle 1 day 8: number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 1 | 2 | 4 | 5 | 3 | 3 | 3 | 1 | 3 | 3 | 5 | 3 | 2 | 4 | 3 | 4 | 4 | 6 | 0 | 0 | 0 | 0 | 9 | 12
  Cycle 1 day 8 | 1740 [1140 to 2930] | 3830 [1660 to 4510] | 3250 [1590 to 4840] | 5650 [3910 to 6470] | 10200 [9740 to 11300] | 39400 [39400 to 39400] | 17700 [10300 to 25000] | 18400 [10600 to 80300] | 18700 [14700 to 22200] | 31900 [28500 to 35300] | 16100 [10600 to 26700] | 15000 [13800 to 17200] | 23800 [23800 to 23800] | 37600 [26700 to 41900] | 5580 [2660 to 12200] | 8500 [6570 to 27200] | 12700 [7140 to 187000] | 12200 [11400 to 12900] | 3770 [2520 to 5420] | 6300 [28.6 to 21300] | 11100 [0.00 to 15100] | 6020 [5730 to 8610] | 1850 [1230 to 18900] |  |  |  |  | 4710 [0.00 to 13500] | 12700 [0.00 to 311000]
  Cycle 1 day 9: number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 1 | 3 | 1 | 5 | 5 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 7
  Cycle 1 day 9 | 2810 [34.7 to 4070] | 3830 [2010 to 6780] | 4480 [824 to 7130] | 6400 [6010 to 7230] | 11400 [11000 to 14100] | 27300 [27300 to 27300] | 15900 [13700 to 29400] | 91100 [91100 to 91100] | 19800 [11900 to 22900] | 21100 [7030 to 21600] |  |  |  |  | 9530 [2700 to 10800] | 8670 [6490 to 10800] | 12100 [7230 to 34900] |  |  |  |  |  |  |  |  |  |  | 6880 [1850 to 26700] | 14300 [40.1 to 52600]
  Cycle 1 day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 2140 [838 to 29300] |  |  |  |  |  |

6. Primary Outcome: Area Under the Concentration-time Curve (AUC) From Time 0 to 24 Hours (AUC0-24) of AMG 176 (Parts 1A, 3A [Cohorts 1, 2, and 3], and 4 [Cohorts 5A and 5B])
Description: Plasma concentrations of AMG 176 were determined using a validated assay. Noncompartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ of 5.00 ng/mL were set to zero before data analysis.
Time Frame: Parts 1A, 3A and, 4: Cycle 1 day 1 pre, EOI, 1, 2, 3, 5, and 7 hrs EOI, cycle 1 day 8 pre and EOI
Population: The PK analysis set included all participants who had received at least 1 dose of AMG 176 and had at least 1 PK sample collected. AUC0-24 was pre-specified in Parts 1A, 3A (Cohorts 1, 2, and 3) and 4 (Cohorts 5A and 5B) and participants with data available at each time point are presented.
Measure: Median (Full Range); unit: hour*ng/mL
Groups:
- Part 3 Cohort 1 (AML): AMG 176 Dose D BIW: Participants with AML received AMG 176 Dose D BIW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 3 Cohort 2 (AML): AMG 176 Dose E BIW: Participants with AML received AMG 176 Dose E BIW. AMG 176 was administered as an IV infusion in a 4-week cycle.
- Part 3 Cohort 3 (AML): AMG 176 Dose E Then Dose F BIW: Participants with AML received AMG 176 Dose E in cycle 1 week 1, then received Dose F BIW. AMG 176 was administered as an IV infusion in a 4-week cycle.
Arm/Group | Part 1A Cohort 1 (MM): AMG 176 Dose A BIW | Part 1A Cohort 2 (MM): AMG 176 Dose B BIW | Part 1A Cohort 3 (MM): AMG 176 Dose C BIW | Part 1A Cohort 4 (MM): AMG 176 Dose D BIW | Part 1A Cohort 5 (MM): AMG 176 Dose E BIW | Part 1A Cohort 6 (MM): AMG 176 Dose G BIW | Part 1A Cohort 7 (MM): AMG 176 Dose E Then Dose F BIW | Part 1A Cohort 8 (MM): AMG 176 Dose E Then Dose G BIW | Part 1A Cohort 9 (MM): AMG 176 Dose E Then Dose H BIW | Part 1A Cohort 10 (MM): AMG 176 Dose E Then Dose I BIW | Part 3 Cohort 1 (AML): AMG 176 Dose D BIW | Part 3 Cohort 2 (AML): AMG 176 Dose E BIW | Part 3 Cohort 3 (AML): AMG 176 Dose E Then Dose F BIW | Part 4 Cohort 5A (AML): AMG 176 Dose E BIW + Azacitidine | Part 4 Cohort 5B (AML): AMG 176 Dose E the Dose G BIW + Azacitidine
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 2 | 3 | 4 | 3 | 2 | 5 | 5 | 3 | 3 | 6
hour*ng/mL
  Cycle 1 day 1: number analyzed (Participants) | 3 | 3 | 4 | 2 | 3 | 0 | 2 | 2 | 2 | 2 | 5 | 5 | 3 | 3 | 5
  Cycle 1 day 1 | 6230 [6100 to 11500] | 13700 [11900 to 16500] | 13900 [3570 to 18700] | 32700 [21300 to 44100] | 48500 [36700 to 60900] |  | 26700 [11000 to 42400] | 128000 [40100 to 216000] | 47700 [38500 to 56800] | 38500 [24100 to 52800] | 18300 [10000 to 28900] | 44700 [17100 to 66100] | 64900 [35900 to 83900] | 30100 [26300 to 50200] | 32000 [22000 to 37100]
  Cycle 1 day 8: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 4 | 3 | 2 | 2 | 5 | 0 | 3 | 6
  Cycle 1 day 8 |  |  | 21100 [21100 to 21100] | 3240 [3240 to 3240] | 130000 [130000 to 130000] |  | 52300 [20600 to 84000] | 128000 [110000 to 345000] | 118000 [111000 to 191000] | 176000 [84600 to 267000] | 52600 [31000 to 74300] | 51800 [48700 to 91300] |  | 23600 [0.00 to 28300] | 86800 [33900 to 133000]

7. Primary Outcome: AUC From Time 0 to 144 Hours (AUC0-144) of AMG 176 (Parts 1A, 3A [Cohorts 1, 2, and 3], and 4 [Cohorts 5A and 5B])
Description: as for outcome 6
Time Frame: Parts 1A, 3A, and 4: Cycle 1 day 2 pre, EOI, 1, 2, 3, 5, and 7 hrs EOI, cycle 1 day 9 pre and EOI
Population: The PK analysis set included all participants who had received at least 1 dose of AMG 176 and had at least 1 PK sample collected. AUC0-144 was pre-specified in Parts 1A, 3A (Cohorts 1, 2, and 3) and 4 (Cohorts 5A and 5B) and participants with data available at each time point are presented.
Measure: Median (Full Range); unit: hour*ng/mL
Arm/Group | Part 1A Cohort 1 (MM): AMG 176 Dose A BIW | Part 1A Cohort 2 (MM): AMG 176 Dose B BIW | Part 1A Cohort 3 (MM): AMG 176 Dose C BIW | Part 1A Cohort 4 (MM): AMG 176 Dose D BIW | Part 1A Cohort 5 (MM): AMG 176 Dose E BIW | Part 1A Cohort 6 (MM): AMG 176 Dose G BIW | Part 1A Cohort 7 (MM): AMG 176 Dose E Then Dose F BIW | Part 1A Cohort 8 (MM): AMG 176 Dose E Then Dose G BIW | Part 1A Cohort 9 (MM): AMG 176 Dose E Then Dose H BIW | Part 1A Cohort 10 (MM): AMG 176 Dose E Then Dose I BIW | Part 3 Cohort 1 (AML): AMG 176 Dose D BIW | Part 3 Cohort 2 (AML): AMG 176 Dose E BIW | Part 3 Cohort 3 (AML): AMG 176 Dose E Then Dose F BIW | Part 4 Cohort 5A (AML): AMG 176 Dose E BIW + Azacitidine | Part 4 Cohort 5B (AML): AMG 176 Dose E the Dose G BIW + Azacitidine
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 0 | 2 | 1 | 2 | 4 | 5 | 5 | 3 | 2 | 6
hour*ng/mL
  Cycle 1 day 2: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 0 | 0 | 1 | 0 | 1 | 5 | 5 | 3 | 2 | 6
  Cycle 1 day 2 | 10800 [8190 to 20000] | 25300 [21100 to 30700] | 25700 [5660 to 33900] | 58900 [45800 to 72000] | 87600 [81200 to 115000] |  |  | 277000 [277000 to 277000] |  | 385000 [385000 to 385000] | 34600 [11500 to 74100] | 81000 [51700 to 173000] | 122000 [51400 to 258000] | 63000 [0.00 to 126000] | 99300 [73600 to 508000]
  Cycle 1 day 9: number analyzed (Participants) | 1 | 3 | 2 | 1 | 2 | 0 | 2 | 1 | 2 | 4 | 2 | 4 | 0 | 1 | 3
  Cycle 1 day 9 | 540000 [540000 to 540000] | 124000 [119000 to 217000] | 234000 [225000 to 242000] | 202000 [202000 to 202000] | 435000 [379000 to 491000] |  | 134000 [20100 to 249000] | 990000 [990000 to 990000] | 518000 [352000 to 684000] | 473000 [293000 to 838000] | 432000 [59100 to 805000] | 197000 [97800 to 313000] |  | 121000 [121000 to 121000] | 217000 [175000 to 284000]

8. Primary Outcome: AUC From Time 0 to 168 Hours (AUC0-168) of AMG 176 (Parts 1B, 3 [Cohort 4], 3B, 3C, and 3D)
Description: as for outcome 6
Time Frame: Parts 1B, 3B, 3C, and 3 (cohort 4): Cycle 1 day 1 pre, EOI, 1, 2, 3, 5, and 7 hrs EOI, cycle 1 day 8 pre, EOI; Part 3d also cycle 1 day 15 pre and EOI
Population: The PK analysis set included all participants who had received at least 1 dose of AMG 176 and had at least 1 PK sample collected. AUC0-168 was pre-specified in Parts 1B, 3 (Cohort 4), 3B, 3C, and 3D and participants with data available at each time point are presented.
Measure: Median (Full Range); unit: hour*ng/mL
Groups:
- Part 3 Cohort 4 (Japanese Participants With AML): AMG 176 Dose E Then Dose F QW: Japanese participants with AML received AMG 176 Dose E in cycle 1 week 1, then received Dose F QW. AMG 176 was administered as an IV infusion in a 4-week cycle.
Arm/Group | Part 1B Cohort 1 (MM): AMG 176 Dose E Then Dose F QW | Part 1B Cohort 2 (MM): AMG 176 Dose E Then Dose G QW | Part 1B Cohort 3 (MM): AMG 176 Dose E Then Dose H QW | Part 1B Cohort 4 (MM): AMG 176 Dose E Then Dose I QW | Part 3 Cohort 4 (Japanese Participants With AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 1 (AML): AMG 176 Dose E QW | Part 3B Cohort 2 (AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 3 (AML): AMG 176 Dose E Then Dose G QW | Part 3C Cohort 1 (Japanese Participants With AML): AMG 176 Dose E QW | Part 3D Cohort 1 (AML): AMG 176 Dose D QW + Itraconazole
Number analyzed (Participants) | 3 | 3 | 1 | 3 | 2 | 4 | 2 | 3 | 4 | 8
hour*ng/mL
  Cycle 1 day 1: number analyzed (Participants) | 3 | 2 | 1 | 2 | 2 | 4 | 2 | 3 | 4 | 8
  Cycle 1 day 1 | 133000 [75600 to 344000] | 152000 [123000 to 181000] | 108000 [108000 to 108000] | 104000 [98300 to 110000] | 199000 [183000 to 214000] | 82200 [76000 to 180000] | 74400 [46800 to 102000] | 83700 [41200 to 106000] | 203000 [138000 to 306000] | 12800 [9390 to 22200]
  Cycle 1 day 8: number analyzed (Participants) | 3 | 3 | 1 | 3 | 2 | 4 | 2 | 3 | 4 | 3
  Cycle 1 day 8 | 185000 [135000 to 271000] | 348000 [309000 to 361000] | 345000 [345000 to 345000] | 405000 [191000 to 1360000] | 296000 [216000 to 376000] | 34800 [21000 to 62300] | 450000 [446000 to 455000] | 272000 [227000 to 619000] | 153000 [65000 to 252000] | 25700 [16600 to 28600]
  Cycle 1 day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Cycle 1 day 15 |  |  |  |  |  |  |  |  |  | 14600 [3530 to 95400]

9. Primary Outcome: Clearance (CL) of AMG 176
Description: Plasma concentrations of AMG 176 were determined using a validated assay. Noncompartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ of 5.00 ng/mL were set to zero before data analysis. Clearance was calculated as Dose/ AUC0-144 for Parts 1A, 3A, and 4; and as Dose/AUC0-168 for Parts 1B, 3 (Cohort 4 only) 3B, 3C, and 3D.
Time Frame: Parts 1B, 3B, 3C, 3A (cohort 4) Cycle 1: day 1 pre, EOI, 1, 2, 3, 5, 7 hrs EOI, day 8 pre, EOI; Part 3D also days 9, 15 pre and EOI; Parts 1A, 3 (except cohort 4), 4: also day 2 pre, EOI, 1, 2, 3, 5, 7 hrs EOI, day 9 pre and EOI
Population: as for outcome 5
Measure: Median (Full Range); unit: mL/hr/m^2
Arm/Group | Part 1A Cohort 1 (MM): AMG 176 Dose A BIW | Part 1A Cohort 2 (MM): AMG 176 Dose B BIW | Part 1A Cohort 3 (MM): AMG 176 Dose C BIW | Part 1A Cohort 4 (MM): AMG 176 Dose D BIW | Part 1A Cohort 5 (MM): AMG 176 Dose E BIW | Part 1A Cohort 6 (MM): AMG 176 Dose G BIW | Part 1A Cohort 7 (MM): AMG 176 Dose E Then Dose F BIW | Part 1A Cohort 8 (MM): AMG 176 Dose E Then Dose G BIW | Part 1A Cohort 9 (MM): AMG 176 Dose E Then Dose H BIW | Part 1A Cohort 10 (MM): AMG 176 Dose E Then Dose I BIW | Part 1B Cohort 1 (MM): AMG 176 Dose E Then Dose F QW | Part 1B Cohort 2 (MM): AMG 176 Dose E Then Dose G QW | Part 1B Cohort 3 (MM): AMG 176 Dose E Then Dose H QW | Part 1B Cohort 4 (MM): AMG 176 Dose E Then Dose I QW | Part 3A Cohort 1 (AML): AMG 176 Dose D BIW | Part 3A Cohort 2 (AML): AMG 176 Dose E BIW | Part 3A Cohort 3 (AML): AMG 176 Dose E Then Dose F BIW | Part 3A Cohort 4 (Japanese Participants With AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 1 (AML): AMG 176 Dose E QW | Part 3B Cohort 2 (AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 3 (AML): AMG 176 Dose E Then Dose G QW | Part 3C Cohort 1 (Japanese Participants With AML): AMG 176 Dose E QW | Part 3D Cohort 1 (AML): AMG 176 Dose D QW + Itraconazole | Part 4 Cohort 1 (AML): AMG 176 Dose D QW + Azacitidine | Part 4 Cohort 2 (AML): AMG 176 Dose E QW + Azacitidine | Part 4 Cohort 3 (AML): AMG 176 Dose E Then Dose F QW + Azacitidine | Part 4 Cohort 4 (AML): AMG 176 Dose E Then Dose G QW + Azacitidine | Part 4 Cohort 5A (AML): AMG 176 Dose E BIW + Azacitidine | Part 4 Cohort 5B (AML): AMG 176 Dose E the Dose G BIW + Azacitidine
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 0 | 2 | 1 | 2 | 3 | 3 | 3 | 1 | 3 | 5 | 5 | 3 | 2 | 4 | 2 | 3 | 4 | 8 | 0 | 0 | 0 | 0 | 1 | 6
mL/hr/m^2
  Cycle 1 day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 2 | 0 | 0 | 0 | 2 | 4 | 2 | 3 | 4 | 8 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 day 1 |  |  |  |  |  |  |  |  |  |  | 0.886 [0.354 to 1.59] | 0.819 [0.670 to 0.968] | 1.17 [1.17 to 1.17] | 1.16 [1.07 to 1.24] |  |  |  | 0.603 [0.556 to 0.650] | 1.47 [0.674 to 1.60] | 1.88 [1.23 to 2.54] | 1.42 [1.14 to 2.82] | 0.605 [0.389 to 0.838] | 4.68 [2.74 to 6.18] |  |  |  |  |  |
  Cycle 1 day 2: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6
  Cycle 1 day 2 | 2.77 [1.50 to 3.66] | 1.58 [1.30 to 1.80] | 1.95 [1.36 to 9.00] | 1.07 [0.834 to 1.31] | 1.36 [1.04 to 1.50] |  |  | 0.430 [0.430 to 0.430] |  | 0.309 [0.309 to 0.309] |  |  |  |  | 1.73 [0.810 to 4.94] | 1.50 [0.698 to 2.28] | 0.981 [0.461 to 2.28] |  |  |  |  |  |  |  |  |  |  | 0.992 [0.992 to 0.992] | 1.20 [0.236 to 1.68]
  Cycle 1 day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 3 | 0 | 0 | 0 | 2 | 4 | 2 | 3 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 day 8 |  |  |  |  |  |  |  |  |  |  | 0.992 [0.664 to 1.31] | 0.686 [0.653 to 0.785] | 1.10 [1.10 to 1.10] | 1.16 [0.357 to 2.57] |  |  |  | 0.652 [0.476 to 0.828] | 3.58 [1.96 to 5.61] | 0.407 [0.391 to 0.422] | 0.854 [0.396 to 1.01] | 0.782 [0.477 to 1.78] | 2.26 [2.10 to 3.62] |  |  |  |  |  |
  Cycle 1 day 9: number analyzed (Participants) | 1 | 3 | 2 | 1 | 2 | 0 | 2 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Cycle 1 day 9 | 0.0556 [0.0556 to 0.0556] | 0.307 [0.185 to 0.335] | 0.218 [0.214 to 0.222] | 0.291 [0.291 to 0.291] | 0.278 [0.243 to 0.314] |  | 4.82 [0.712 to 8.93] | 0.242 [0.242 to 0.242] | 0.756 [0.513 to 1.000] | 1.14 [0.560 to 1.65] |  |  |  |  | 0.544 [0.0733 to 1.01] | 0.744 [0.393 to 1.24] |  |  |  |  |  |  |  |  |  |  |  | 0.978 [0.978 to 0.978] | 1.11 [0.856 to 1.36]
  Cycle 1 day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 4.08 [0.640 to 15.9] |  |  |  |  |  |

10. Primary Outcome: Terminal Half-life (t1/2) of AMG 176
Description: as for outcome 6
Time Frame: as for outcome 9
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1A Cohort 1 (MM): AMG 176 Dose A BIW | Part 1A Cohort 2 (MM): AMG 176 Dose B BIW | Part 1A Cohort 3 (MM): AMG 176 Dose C BIW | Part 1A Cohort 4 (MM): AMG 176 Dose D BIW | Part 1A Cohort 5 (MM): AMG 176 Dose E BIW | Part 1A Cohort 6 (MM): AMG 176 Dose G BIW | Part 1A Cohort 7 (MM): AMG 176 Dose E Then Dose F BIW | Part 1A Cohort 8 (MM): AMG 176 Dose E Then Dose G BIW | Part 1A Cohort 9 (MM): AMG 176 Dose E Then Dose H BIW | Part 1A Cohort 10 (MM): AMG 176 Dose E Then Dose I BIW | Part 1B Cohort 1 (MM): AMG 176 Dose E Then Dose F QW | Part 1B Cohort 2 (MM): AMG 176 Dose E Then Dose G QW | Part 1B Cohort 3 (MM): AMG 176 Dose E Then Dose H QW | Part 1B Cohort 4 (MM): AMG 176 Dose E Then Dose I QW | Part 3A Cohort 1 (AML): AMG 176 Dose D BIW | Part 3A Cohort 2 (AML): AMG 176 Dose E BIW | Part 3A Cohort 3 (AML): AMG 176 Dose E Then Dose F BIW | Part 3A Cohort 4 (Japanese Participants With AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 1 (AML): AMG 176 Dose E QW | Part 3B Cohort 2 (AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 3 (AML): AMG 176 Dose E Then Dose G QW | Part 3C Cohort 1 (Japanese Participants With AML): AMG 176 Dose E QW | Part 3D Cohort 1 (AML): AMG 176 Dose D QW + Itraconazole | Part 4 Cohort 1 (AML): AMG 176 Dose D QW + Azacitidine | Part 4 Cohort 2 (AML): AMG 176 Dose E QW + Azacitidine | Part 4 Cohort 3 (AML): AMG 176 Dose E Then Dose F QW + Azacitidine | Part 4 Cohort 4 (AML): AMG 176 Dose E Then Dose G QW + Azacitidine | Part 4 Cohort 5A (AML): AMG 176 Dose E BIW + Azacitidine | Part 4 Cohort 5B (AML): AMG 176 Dose E the Dose G BIW + Azacitidine
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 1 | 1 | 1 | 3 | 3 | 1 | 2 | 0 | 1 | 5 | 4 | 4 | 0 | 1 | 2 | 2 | 1 | 5 | 0 | 0 | 0 | 0 | 2 | 5
hours
  Cycle 1 day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 day 1 |  |  |  |  |  |  |  |  |  |  | 19.6 [19.6 to 19.6] |  |  | 2.58 [2.58 to 2.58] |  |  |  |  | 2.62 [2.62 to 2.62] |  | 47.3 [47.3 to 47.3] | 17.4 [17.4 to 17.4] | 4.42 [2.91 to 10.2] |  |  |  |  |  |
  Cycle 1 day 2: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5
  Cycle 1 day 2 | 3.33 [2.46 to 8.20] | 9.18 [6.93 to 9.55] | 7.66 [3.14 to 10.7] | 7.98 [7.34 to 8.61] | 7.43 [6.31 to 10.4] | 11.3 [11.3 to 11.3] |  | 18.5 [18.5 to 18.5] |  |  |  |  |  |  | 15.3 [3.63 to 58.9] | 20.6 [5.69 to 33.6] | 6.85 [5.04 to 19.3] |  |  |  |  |  |  |  |  |  |  | 17.7 [5.78 to 29.6] | 9.98 [7.44 to 24.3]
  Cycle 1 day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 day 8 |  |  |  |  |  |  |  |  |  |  |  | 46.7 [25.6 to 67.7] |  | 28.3 [28.3 to 28.3] |  |  |  |  | 3.70 [3.70 to 3.70] | 35.6 [30.8 to 40.4] | 11.7 [5.44 to 18.1] | 17.8 [17.8 to 17.8] |  |  |  |  |  |  |
  Cycle 1 day 9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
  Cycle 1 day 9 |  |  |  |  |  |  | 1.05 [1.05 to 1.05] | 44.5 [44.5 to 44.5] | 12.9 [10.9 to 14.6] | 16.9 [12.6 to 20.5] |  |  |  |  | 34.0 [34.0 to 34.0] | 24.6 [21.9 to 42.0] | 9.81 [8.17 to 11.5] |  |  |  |  |  |  |  |  |  |  | 4.33 [4.08 to 4.59] | 15.4 [7.06 to 17.3]
  Cycle 1 day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 9.08 [9.08 to 9.08] |  |  |  |  |  |

ADVERSE EVENTS:
Time Frame: For mortality, from enrolment to end of study; median time on study was 2.3 months. For AEs, from first dose of AMG 176 to 30 days after the last dose of AMG 176; median treatment duration was 1.2 months.
Groups:
- Part 4 Cohort 2 (AML): AMG 176 Dose E QW + Azacitidine: Participants with AML received AMG 176 Dose E QW. AMG 176 was administered as an IV infusion in a 4-week cycle. They also received 75 mg/m^2 azacitidine SC or IV QD for the first 7 days of the 4-week cycle.
Arm/Group | Part 1A Cohort 1 (MM): AMG 176 Dose A BIW | Part 1A Cohort 2 (MM): AMG 176 Dose B BIW | Part 1A Cohort 3 (MM): AMG 176 Dose C BIW | Part 1A Cohort 4 (MM): AMG 176 Dose D BIW | Part 1A Cohort 5 (MM): AMG 176 Dose E BIW | Part 1A Cohort 6 (MM): AMG 176 Dose G BIW | Part 1A Cohort 7 (MM): AMG 176 Dose E Then Dose F BIW | Part 1A Cohort 8 (MM): AMG 176 Dose E Then Dose G BIW | Part 1A Cohort 9 (MM): AMG 176 Dose E Then Dose H BIW | Part 1A Cohort 10 (MM): AMG 176 Dose E Then Dose I BIW | Part 1B Cohort 1 (MM): AMG 176 Dose E Then Dose F QW | Part 1B Cohort 2 (MM): AMG 176 Dose E Then Dose G QW | Part 1B Cohort 3 (MM): AMG 176 Dose E Then Dose H QW | Part 1B Cohort 4 (MM): AMG 176 Dose E Then Dose I QW | Part 3A Cohort 1 (AML): AMG 176 Dose D BIW | Part 3A Cohort 2 (AML): AMG 176 Dose E BIW | Part 3A Cohort 3 (AML): AMG 176 Dose E Then Dose F BIW | Part 3A Cohort 4 (Japanese Participants With AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 1 (AML): AMG 176 Dose E QW | Part 3B Cohort 2 (AML): AMG 176 Dose E Then Dose F QW | Part 3B Cohort 3 (AML): AMG 176 Dose E Then Dose G QW | Part 3C Cohort 1 (Japanese Participants With AML): AMG 176 Dose E QW | Part 3D Cohort 1 (AML): AMG 176 Dose D QW + Itraconazole | Part 4 Cohort 1 (AML): AMG 176 Dose D QW + Azacitidine | Part 4 Cohort 2 (AML): AMG 176 Dose E QW + Azacitidine | Part 4 Cohort 3 (AML): AMG 176 Dose E Then Dose F QW + Azacitidine | Part 4 Cohort 4 (AML): AMG 176 Dose E Then Dose G QW + Azacitidine | Part 4 Cohort 5A (AML): AMG 176 Dose E BIW + Azacitidine | Part 4 Cohort 5B (AML): AMG 176 Dose E the Dose G BIW + Azacitidine
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/4 | 0/3 | 0/3 | 1/2 | 0/4 | 0/4 | 1/5 | 0/5 | 0/3 | 0/3 | 1/3 | 0/3 | 0/5 | 2/5 | 0/5 | 0/2 | 4/4 | 3/3 | 3/4 | 3/4 | 7/10 | 5/5 | 3/4 | 4/4 | 7/13 | 6/10 | 9/13
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/4 | 0/3 | 1/3 | 2/2 | 3/4 | 0/4 | 2/5 | 3/5 | 0/3 | 2/3 | 1/3 | 1/3 | 3/5 | 4/5 | 3/5 | 2/2 | 2/4 | 2/3 | 4/4 | 1/4 | 8/10 | 4/5 | 4/4 | 4/4 | 10/13 | 8/10 | 10/13
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 4/4 | 3/3 | 3/3 | 1/2 | 4/4 | 4/4 | 5/5 | 5/5 | 3/3 | 3/3 | 3/3 | 3/3 | 4/5 | 3/5 | 5/5 | 2/2 | 4/4 | 3/3 | 4/4 | 4/4 | 10/10 | 5/5 | 4/4 | 4/4 | 13/13 | 10/10 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A Cohort 1 (MM): AMG 176 Dose A BIW (N=3) | Part 1A Cohort 2 (MM): AMG 176 Dose B BIW (N=3) | Part 1A Cohort 3 (MM): AMG 176 Dose C BIW (N=4) | Part 1A Cohort 4 (MM): AMG 176 Dose D BIW (N=3) | Part 1A Cohort 5 (MM): AMG 176 Dose E BIW (N=3) | Part 1A Cohort 6 (MM): AMG 176 Dose G BIW (N=2) | Part 1A Cohort 7 (MM): AMG 176 Dose E Then Dose F BIW (N=4) | Part 1A Cohort 8 (MM): AMG 176 Dose E Then Dose G BIW (N=4) | Part 1A Cohort 9 (MM): AMG 176 Dose E Then Dose H BIW (N=5) | Part 1A Cohort 10 (MM): AMG 176 Dose E Then Dose I BIW (N=5) | Part 1B Cohort 1 (MM): AMG 176 Dose E Then Dose F QW (N=3) | Part 1B Cohort 2 (MM): AMG 176 Dose E Then Dose G QW (N=3) | Part 1B Cohort 3 (MM): AMG 176 Dose E Then Dose H QW (N=3) | Part 1B Cohort 4 (MM): AMG 176 Dose E Then Dose I QW (N=3) | Part 3A Cohort 1 (AML): AMG 176 Dose D BIW (N=5) | Part 3A Cohort 2 (AML): AMG 176 Dose E BIW (N=5) | Part 3A Cohort 3 (AML): AMG 176 Dose E Then Dose F BIW (N=5) | Part 3A Cohort 4 (Japanese Participants With AML): AMG 176 Dose E Then Dose F QW (N=2) | Part 3B Cohort 1 (AML): AMG 176 Dose E QW (N=4) | Part 3B Cohort 2 (AML): AMG 176 Dose E Then Dose F QW (N=3) | Part 3B Cohort 3 (AML): AMG 176 Dose E Then Dose G QW (N=4) | Part 3C Cohort 1 (Japanese Participants With AML): AMG 176 Dose E QW (N=4) | Part 3D Cohort 1 (AML): AMG 176 Dose D QW + Itraconazole (N=10) | Part 4 Cohort 1 (AML): AMG 176 Dose D QW + Azacitidine (N=5) | Part 4 Cohort 2 (AML): AMG 176 Dose E QW + Azacitidine (N=4) | Part 4 Cohort 3 (AML): AMG 176 Dose E Then Dose F QW + Azacitidine (N=4) | Part 4 Cohort 4 (AML): AMG 176 Dose E Then Dose G QW + Azacitidine (N=13) | Part 4 Cohort 5A (AML): AMG 176 Dose E BIW + Azacitidine (N=10) | Part 4 Cohort 5B (AML): AMG 176 Dose E the Dose G BIW + Azacitidine (N=13)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 3 | 2 | 3 | 4 | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric mucosal lesion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemophilus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 5 | 4 | 5
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 2 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Superinfection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
JC polyomavirus test (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laboratory test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial necrosis marker increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A Cohort 1 (MM): AMG 176 Dose A BIW (N=3) | Part 1A Cohort 2 (MM): AMG 176 Dose B BIW (N=3) | Part 1A Cohort 3 (MM): AMG 176 Dose C BIW (N=4) | Part 1A Cohort 4 (MM): AMG 176 Dose D BIW (N=3) | Part 1A Cohort 5 (MM): AMG 176 Dose E BIW (N=3) | Part 1A Cohort 6 (MM): AMG 176 Dose G BIW (N=2) | Part 1A Cohort 7 (MM): AMG 176 Dose E Then Dose F BIW (N=4) | Part 1A Cohort 8 (MM): AMG 176 Dose E Then Dose G BIW (N=4) | Part 1A Cohort 9 (MM): AMG 176 Dose E Then Dose H BIW (N=5) | Part 1A Cohort 10 (MM): AMG 176 Dose E Then Dose I BIW (N=5) | Part 1B Cohort 1 (MM): AMG 176 Dose E Then Dose F QW (N=3) | Part 1B Cohort 2 (MM): AMG 176 Dose E Then Dose G QW (N=3) | Part 1B Cohort 3 (MM): AMG 176 Dose E Then Dose H QW (N=3) | Part 1B Cohort 4 (MM): AMG 176 Dose E Then Dose I QW (N=3) | Part 3A Cohort 1 (AML): AMG 176 Dose D BIW (N=5) | Part 3A Cohort 2 (AML): AMG 176 Dose E BIW (N=5) | Part 3A Cohort 3 (AML): AMG 176 Dose E Then Dose F BIW (N=5) | Part 3A Cohort 4 (Japanese Participants With AML): AMG 176 Dose E Then Dose F QW (N=2) | Part 3B Cohort 1 (AML): AMG 176 Dose E QW (N=4) | Part 3B Cohort 2 (AML): AMG 176 Dose E Then Dose F QW (N=3) | Part 3B Cohort 3 (AML): AMG 176 Dose E Then Dose G QW (N=4) | Part 3C Cohort 1 (Japanese Participants With AML): AMG 176 Dose E QW (N=4) | Part 3D Cohort 1 (AML): AMG 176 Dose D QW + Itraconazole (N=10) | Part 4 Cohort 1 (AML): AMG 176 Dose D QW + Azacitidine (N=5) | Part 4 Cohort 2 (AML): AMG 176 Dose E QW + Azacitidine (N=4) | Part 4 Cohort 3 (AML): AMG 176 Dose E Then Dose F QW + Azacitidine (N=4) | Part 4 Cohort 4 (AML): AMG 176 Dose E Then Dose G QW + Azacitidine (N=13) | Part 4 Cohort 5A (AML): AMG 176 Dose E BIW + Azacitidine (N=10) | Part 4 Cohort 5B (AML): AMG 176 Dose E the Dose G BIW + Azacitidine (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 1 | 3 | 4 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0
Coagulation factor deficiency (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 2 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 4 | 1 | 3 | 2 | 2 | 1 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stress polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 2
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chondrodermatitis nodularis chronica helicis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conductive deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mastoid effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eczema eyelids (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scleral disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scleral haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 2 | 4
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 4 | 4 | 1 | 3 | 2 | 2 | 1 | 1 | 1 | 0 | 2 | 2 | 2 | 0 | 3 | 3 | 1 | 3 | 7 | 7 | 6
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 0 | 1 | 3 | 1 | 4 | 3 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 2 | 2 | 1 | 3 | 3 | 3 | 2 | 7 | 8 | 6
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral blood blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Oral purpura (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tongue haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Traumatic occlusion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 5 | 1 | 1 | 2 | 3 | 3 | 0 | 2 | 1 | 1 | 3 | 2 | 0 | 2 | 3 | 1 | 2 | 7 | 5 | 3
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 2
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 1 | 5 | 3 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 4 | 2 | 2 | 0 | 2 | 2 | 5
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site irritation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site phlebitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Injection site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Non-pitting oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 1 | 3 | 2 | 1 | 0 | 1 | 1 | 0 | 3 | 3 | 0 | 1 | 4 | 3 | 2
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 3 | 1 | 1
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periportal oedema (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Citrobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pertussis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 3
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 3
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2
Aspartate aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 5
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile acids increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Biopsy skin normal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blast cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0
Blood lactate dehydrogenase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
CSF white blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haptoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 3 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 3
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pulmonary arterial pressure abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory syncytial virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respirovirus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 3 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 3 | 4 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 4 | 2 | 0 | 1 | 5 | 4 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 2 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 2 | 1 | 0 | 1 | 1 | 4
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight fluctuation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 2 | 3
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 0 | 2 | 5 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyporeflexia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Frustration tolerance decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnambulism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 2 | 1 | 0 | 3 | 3 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 1 | 3 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 3 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 2 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Debridement (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Knee operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aortic dilatation (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arterial disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 3 | 1 | 3
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular pain (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was conducted in multiple parts and Part 5 did not enroll any participants due to early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT02675452/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT02675452/SAP_001.pdf